CLINICAL TRIAL: NCT06924476
Title: Optimization of a Decision Formula for Optimal Timing of Immunosuppressive Therapy Initiation in Primary Membranous Nephropathy: A Multicenter Retrospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Yipeng Liu (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(064)
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Primary Membranous Nephropathy
Keywords: Primary Membranous Nephropathy; Evaluation formula; Initiate immunosuppressive therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modeling Group: The data of this group of participants are used to construct the evaluation formula.
- Verification group: The data of this group of participants are used to verify the evaluation formula constructed through the modeling group.

SUMMARY:
The goal of this observational study is to optimize the evaluation formula for the timing of initiating immunosuppressive therapy in primary membranous nephropathy in patients with primary membranous nephropathy. The main question it aims to answer is:When should immunosuppressive therapy be initiated?This study is a retrospective one. Participants will not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* It meets one of the diagnostic criteria for PMN as stipulated in the KDIGO 2021 Clinical Practice Guidelines for the Management of Glomerular Diseases: patients with a clear diagnosis of PMN based on renal biopsy pathology or presenting with nephrotic syndrome and positive anti-PLA2R antibody detection (>14RU/mL), and excluding secondary factors such as tumors, infections, drugs, and systemic autoimmune diseases.

Exclusion Criteria:

* (1) Patients who have received treatment with immunosuppressive medications other than oral prednisolone.

  (2) The time interval between the renal biopsy and the baseline measurement is longer than 3 years.

  (3) Initiate the use of immunosuppressive agents within 1 week after the diagnosis of PMN.

  (4) Participate in the immunosuppressive treatment trial during the follow-up period and be in the intervention group.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were registered in the Renal Disease Syndrome Multi-center Cohort Network (https://nsn.bjmu.edu.cn/index) and whose medical records were complete, and who met the PMN diagnostic criteria as stipulated in the KDIGO 2021 Clinical Practice Guidelines for the Management of Glomerular Diseases.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 1990-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reasonably add immunosuppressive therapy | From enrollment to the reasonable addition of immunosuppressive agent treatme，no less than one weeknt
  Reasonably add immunosuppressive therapy, that is, refer to the risk stratification of PMN in the "KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases". Immunosuppressive therapy can be initiated for patients with moderate or higher risk; or for those whom the treating doctor deems to require immunosuppressive therapy due to severe and incurable nephrotic syndrome and its serious complications. Meeting either of the two conditions is sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Yipeng Liu, Study Chair — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No